CLINICAL TRIAL: NCT05146115
Title: Validity and Reliability of the Modified Athletic Shoulder Test
Brief Title: Validation of Modified AST
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Camille Tooth, Physiotherapist, University of Liege
Other Study IDs: modified AST
Record Dates: First submitted 2021-11-02; First posted 2021-12-06 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Realization of the Athletic Shoulder Test and the Modified Athletic Shoulder Test — The participants will have to perform both tests two times, with a 7-10 days rest period between the two sessions

SUMMARY:
The objective of the study is the validate and to assess the reliability of a modified version of the Athetic Shoulder Test. The activity of peri-scapular muscles during the realization of the test will be assessed too.

DETAILED DESCRIPTION:
The study will be divided into two sessions. A time of 7-10 days will be provided between the two sessions of tests to limit the influence of sport and training on the results.

Session 1:

* Warm-up
* Realization of the Athletic Shoulder Test (with EMG captors on upper trapezius, lower trapezius and serratus anterior)
* Realization of the modified Athletic Shoulder Test (with EMG captors on upper trapezius, lower trapezius and serratus anterior)

Session 2:

* Warm-up
* Realization of the Athletic Shoulder Test (with EMG captors on upper trapezius, lower trapezius and serratus anterior)
* Realization of the modified Athletic Shoulder Test (with EMG captors on upper trapezius, lower trapezius and serratus anterior)

ELIGIBILITY:
Inclusion Criteria:

* to practice an overhead sport at least 5 hours a week

Exclusion Criteria:

* no shoulder pain
* no history of shoulder pain
* no history of shoulder surgery
* no scoliosis or lower limb lengths differences

Ages: 18 Years to 35 Years | Sex: Male
Age Groups: Adult
Study Population: The participants will have to practice an overhead sport at least 5 hours a week
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Strength of anteflexors in "I" position | Change from baseline to 10 days
  The strength developped in the "I" position will be assessed with a force plateform and a handheld dynamometer
Strength of anteflexors in "Y" position | Change from baseline to 10 days
  The strength developped in the "Y" position will be assessed with a force plateform and a handheld dynamometer
Strength of anteflexors in "T" position | Change from baseline to 10 days
  The strength developped in "T" position will be assessed with a force plateform and a handheld dynamometer
EMG activity of upper trapezius | during the first session
  EMG activity of upper trapezius will be measured with surface electrodes (Delsys Trigno)
EMG activity of lower trapezius | during the first session
  EMG activity of lower trapezius will be measured with surface electrodes (Delsys Trigno)
EMG activity of serratus anterior | during the first session
  EMG activity of serratus anterior will be measured with surface electrodes (Delsys Trigno)

CONTACTS AND LOCATIONS:
Overall Officials: Camille Tooth, Principal Investigator — ULiège
Locations (1):
- Laboratoire d'Analyse du Mouvement Humain, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No